CLINICAL TRIAL: NCT04848168
Title: Comparison Of PRISM III, PIM2 And PELOD Scoring Systems In Predicting Mortality For Patients Undergoing Congenital Cardiac Surgery In Pediatric Intensive Care Unit
Brief Title: Comparison of PRISM III, PIM2 and PELOD Scoring Systems
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Collaborators: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other); Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyma Sayit, principal investigator, Haydarpasa Numune Training and Research Hospital
Other Study IDs: Dr. Siyami Ersek TRH
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Congenital Heart Disease
Keywords: PRISM III; PIM2; PELOD; STAT; mortality; congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PRISMIII(Pediatric Risk of Mortality III), PIM2(Pediatric Index of Mortality 2) and PELOD(Pediatric Logistic Organ Dysfunction) are frequently used for predicting mortality and morbidity in general pediatric ICUs(Intensive Care Units). However, the effectiveness of these scoring sistems in a specific group patients undergoing congenital heart surgery(CHS) is unknown. In this study, the investigators aimed primarily to evaluate the success of these scoring systems in predicting mortality and morbiditiy in this specific group and to compare the scoring systems with eachother, and secondly to evaluate the relationship of these systems with the STAT(STS-EACTS CHS Mortality Score) category

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 18 years of age who had undergone congenital heart surgery

Exclusion Criteria:

* emergency operations Patients staying in intensive care unit for less than 24 hours

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients younger than 18 years of age who had undergone congenital heart surgery
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
evaluate the success of PRISMIII, PIM2 and PELOD scoring systems in predicting mortality and morbidity | 3 months
  Patients younger than 18 years of age who had undergone congenital heart surgery were evaluated on the first postoperative day in the ICU and parameters were recorded. PRISMIII and PELOD scores were calculated using the most abnormal values in the first 24 hours, and PIM2 score was calculated using the data within the first hour.
morbidity indicators | 3 months
  Morbidity indicators were determined as the length of ICU stay, total hospital stay, re-intubation, surgical revision, complications and re-admission to the ICU.
clinical outcomes | 3 months
  Clinical outcomes were determined as 7-day mortality and 30-day mortality.

SECONDARY OUTCOMES:
to evaluate the relationship of these systems with the STAT(STS-EACTS CHS Mortality Score) category | 3 months
  STAT category was determined according to the surgical procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- siyami ersek TRH, Istanbul, Turkey (Türkiye)